CLINICAL TRIAL: NCT05282316
Title: Impact of Extra Virgin Olive Oil (EVOO) with Health Properties in Improving the Overall Health Status and Preventing Cardiovascular Risk in Metabolic Syndrome
Brief Title: Impact of Extra Virgin Olive Oil (EVOO) with Health Properties in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Aurelio Seidita, Research Fellow, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASMS01
Record Dates: First submitted 2022-02-18; First posted 2022-03-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Syndrome
Keywords: Extra Virgin Olive Oil (EVOO); Metabolic syndrome; Mediterranean diet; Polyphenols; Cardiovascular risk; Liver steatosis; Inflammation
MeSH Terms: conditions — Metabolic Syndrome; Fatty Liver; Inflammation

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Same organoleptic features of the two different kind of EVOO (polyphenols enriched and standard).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EVOO polyphenols enriched (Active Comparator): Fifteen subjects with metabolic syndrome will be randomly enrolled each year (3 years of study planned), to the addition of 40 ml daily of healthy polyphenols enriched EVOO to their mediterranean diet for the duration of six months
  Interventions: Dietary Supplement: EVOO polyphenols enriched
- EVOO standard (Placebo Comparator): Fifteen subjects with metabolic syndrome will be randomly enrolled each year (3 years of study planned), to the addition of 40 ml daily of standard EVOO to their mediterranean diet for the duration of six months
  Interventions: Dietary Supplement: EVOO standard

INTERVENTIONS:
Dietary Supplement: EVOO polyphenols enriched — Addition of 40 ml daily of healthy polyphenols enriched EVOO to mediterranean diet for 6 months
  Arms: EVOO polyphenols enriched
Dietary Supplement: EVOO standard — Addition of 40 ml daily of standard EVOO to mediterranean diet for 6 months
  Arms: EVOO standard

SUMMARY:
Metabolic syndrome (MS), defined according to the revised Adult Treatment Panel III - National Cholesterol Education Program (ATP III - NCEP) criteria, represents a widespread condition in Western populations (prevalence ranging from 22% to about 33%) and with a trend that increases with time and age. MS, not differently from each of the components that characterize it, is a known risk factor for cardiovascular and metabolic diseases. To date, national and international panels indicate lifestyle modification as the only indication for treating MS and reducing the risk of cardiovascular and metabolic diseases. The increase in daily physical activity and the modification of the diet are therefore the cornerstones of the treatment.

The Mediterranean Diet (MD) represents a traditional value of the Italian population which has shown in several studies a protective effect on mortality and survival free from cardiovascular events. The added value of MD is the presence of extra virgin olive oil (EVOO), a healthy food with high content of monounsaturated fatty acids, especially oleic acid, and variable concentrations (range 50-800 mg/kg) of phenols (oleuropein, ligstroside, and oleocanthal, and their derivatives phenolic alcohols, such as hydroxytyrosol and tyrosol). Olive oil is defined as healthy according to EC Reg. 432/2012. A good EVOO contains about 75% of oleic acid although a variability between 55% and 83% of all fatty acids is expected according to the World Health Organization. The polyphenols content plays a key role in the choice of the type and quantity of oil with health objectives, with particular reference to the unsaturated and polyunsaturated component (oleic acid, linoleic acid, alpha linolenic acid). Phenolic compounds not only determine EVOO main organoleptic qualities (oxidative stability and specific flavor and taste features) but, theoretically, make it a substance with antioxidant, antiinflammatory, insulin-sensitizing, cardioprotective, antiatherogenic, neuroprotective, immunomodulatory and anticancer activity.

The study aims to use a polyphenols enriched EVOO with health properties, derived from different cultivation variants of olives (cultivars), chosen on the basis of preliminary research, coming from Sicilian harvesting campaigns, to evaluate its potential to modify 'in vivo', in subjects with MS, some clinical and laboratory parameters inferring cardiovascular risk, metabolism and inflammation.

DETAILED DESCRIPTION:
Metabolic syndrome (MS), defined according to the to the revised Adult Treatment Panel III - National Cholesterol Education Program (ATP III - NCEP) criteria,, represents a widespread condition in Western populations (absolute prevalence ranging from 22% to about 33%) and with a trend that increases with time and age (it is expected that its prevalence will increase by about 53% by 2035). MS, not differently from each of the components that characterize it, is a known risk factor for cardiovascular diseases (relative risk (RR) 1.53-2.18) and type 2 diabetes mellitus (RR 3.53-5.17). To date, national and international panels indicate lifestyle modification as the only indication for treating MS and reducing the risk of cardiovascular and metabolic diseases. The increase in daily physical activity and the modification of the diet are therefore the cornerstones of the treatment.

The Mediterranean Diet (MD) represents a traditional value of the Italian population which has shown in several studies a protective effect on mortality and survival free from cardiovascular events. The added value of MD is the presence of extra virgin olive oil (EVOO), a healthy food with high content of monounsaturated fatty acids, especially oleic acid, and variable concentrations (range 50-800 mg/kg) of phenols (oleuropein, ligstroside, and oleocanthal, and their derivatives phenolic alcohols, such as hydroxytyrosol and tyrosol). Olive oil is defined as healthy according to European Commission (EC) Reg. 432/2012. A good EVOO contains about 75% of oleic acid although a variability between 55% and 83% of all fatty acids is expected according to the World Health Organization. The polyphenols content plays a key role in the choice of the type and quantity of oil with health objectives, with particular reference to the unsaturated and polyunsaturated component (oleic acid, linoleic acid, alpha linolenic acid). Phenolic compounds not only determine EVOO main organoleptic qualities (oxidative stability and specific flavor and taste features) but, theoretically, make it a substance with antioxidant, antiinflammatory, insulin-sensitizing, cardioprotective, antiatherogenic, neuroprotective, immunomodulatory and anticancer activity.

Any beneficial substance, including olive oil, goes through a series of biochemical processes before reaching the target organ, by the digestive enzymes and bacteria of the gut microbiota, or the eventual formation of active metabolites after the first liver passage; thus, an exclusively 'in vitro' evaluation of a substance on target cells does not always represent the physiological model of the interaction of these substances with the organism.

The study aims to use a polyphenols enriched EVOO with health properties, derived from different cultivation variants of olives (cultivars), chosen on the basis of preliminary research, coming from Sicilian harvesting campaigns, to evaluate its potential to modify 'in vivo', in subjects with MS, some clinical and laboratory parameters inferring cardiovascular risk, metabolism and inflammation.

Preliminarily, in the phase of the olive harvesting campaigns (three different harvesting periods carried out between November and December: green, mature and advanced ripening), the different indigenous cultivars coming from the same area of Western Sicily (precisely from Val di Mazara, Valle del Belice, Trapani valleys and called Biancolilla, Nocellara, Cerasuolo) will be subjected to biochemical analyses which will aim to identify those with the highest oleic acid and polyphenols content, which will contribute to the enhancement of the specific territory and to the maintenance of biodiversity.

The general objective of the study is to strengthen and enhance the research chain in the nutraceutical and health food sector and the cooperation between the research system and local companies, to support the maximum diffusion and use of new therapeutic substances and advanced technologies for treatment and prevention, and, at the same time, contributing to competitiveness and economic growth by raising the level of scientific-technical skills and knowledge in the production system and in Institutions.

The main objectives of the research, therefore, will be the following:

1. Identification and selection of specific autochthonous cultivar able to provide a high quality and polyphenols enriched EVOO.
2. Establish potential benefits of a polyphenols enriched EVOO-MD assessing the improvement over metabolic (lipidic and glycemic status), inflammatory (cytokines) and cardiovascular (cIMT and endothelial dysfunction) parameters.
3. Establish potential benefits of a polyphenols enriched EVOO-MD assessing the improvement over liver steatosis.
4. Analysis of polyphenols enriched EVOO effects on peripheral blood mononuclear cells (PBMC) gene expression exploring their potential use as diagnostic and therapeutic response tool.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of metabolic syndrome according the revised NCEP ATP III criteria; three or more of the following five criteria are met: waist circumference over 102 cm/40 inches (men) or 88 cm/35 inches (women), blood pressure over 130/85 mmHg, fasting triglyceride level over 150 mg/dl, fasting high-density lipoprotein cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women) and fasting blood sugar over 100 mg/dl.
* Hepatitis B virus (HBV) and hepatitis C virus (HCV) negativity.

Exclusion Criteria:

* alcohol intake (>30 g/day for men and >20 g/day for women);
* acute or chronic hepatic and/or cardiac failure;
* acute or chronic kidney disease (stage G4 Kidney Disease: Improving Global Outcomes (KDIGO) revised classification, glomerular filtration rate <30 mL/min/1.73 m2);
* neoplasms;
* autoimmune or acute and chronic inflammatory diseases;
* acute or chronic infective diseases;
* pregnancy and/or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Change of glycemic control induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p<0.05) from baseline (T0) to end of intervention (T1) of glycated hemoglobin levels.
Change of insulin resistance induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p<0.05) from baseline (T0) to end of intervention (T1) of (HOMA-IR) index.
Change of high density lipoproteins levels induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p<0.05) from baseline (T0) to end of intervention (T1) of high density lipoproteins (HDL) levels.
Change of triglycerides levels induced by polyphenols enriched | From baseline to end of intervention (6 months)
  Statistically significant change (p<0.05) from baseline (T0) to end of intervention (T1) of triglycerides levels.
Change of inflammatory parameter tumor necrosis factor (TNF)-α induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p<0.05) from baseline (T0) to end of intervention (T1) of TNF-α levels.
Change of inflammatory parameter interleukine (IL)-6, induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p<0.05) from baseline (T0) to end of intervention (T1) of tumor necrosis factor IL-6 levels.

SECONDARY OUTCOMES:
Change in liver steatosis ultrasound pattern induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change from baseline (T0) to end of intervention (T1) of liver ultrasound steatosis pattern by ultrasonography.
Change in visceral fat thickness induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p<0.05) from baseline (T0) to end of intervention (T1) of visceral fat thickness by ultrasonography.
Change in carotid intima-media thickness (cIMT) induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p <0.05) from baseline (T0) to end of intervention (T1) of cIMT by ultrasonography.
Change in endothelial disfunction induced by polyphenols enriched EVOO-MD. | From baseline to end of intervention (6 months)
  Statistically significant change (p <0.05) from baseline (T0) to end of intervention (T1) in endothelial dysfunction, by flow-mediated dilatation technique of the brachial artery.
EVOO effects on PBMC stress response gene expression | From baseline to end of intervention (6 months)
  Statistically significant change (p <0.05) from baseline (T0) to end of intervention (T1) of expression of nuclear protein 1 (NUPR1)
EVOO effects on PBMC lipid metabolism gene expression | From baseline to end of intervention (6 months)
  Statistically significant change (p <0.05) from baseline (T0) to end of intervention (T1) of expression of Acetyl-Coenzyme A Carboxylase 1 (ACC1).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Soresi, MD, Study Director — maurizio.soresi@unipa.it
Locations (1):
- Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Costa F; American Heart Association; National Heart, Lung, and Blood Institute. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute Scientific Statement. Circulation. 2005 Oct 25;112(17):2735-52. doi: 10.1161/CIRCULATIONAHA.105.169404. Epub 2005 Sep 12. No abstract available. PMID 16157765
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Pastor R, Bouzas C, Tur JA. Beneficial effects of dietary supplementation with olive oil, oleic acid, or hydroxytyrosol in metabolic syndrome: Systematic review and meta-analysis. Free Radic Biol Med. 2021 Aug 20;172:372-385. doi: 10.1016/j.freeradbiomed.2021.06.017. Epub 2021 Jun 18. PMID 34153478
- [Background] Schwingshackl L, Christoph M, Hoffmann G. Effects of Olive Oil on Markers of Inflammation and Endothelial Function-A Systematic Review and Meta-Analysis. Nutrients. 2015 Sep 11;7(9):7651-75. doi: 10.3390/nu7095356. PMID 26378571
- [Background] George ES, Marshall S, Mayr HL, Trakman GL, Tatucu-Babet OA, Lassemillante AM, Bramley A, Reddy AJ, Forsyth A, Tierney AC, Thomas CJ, Itsiopoulos C, Marx W. The effect of high-polyphenol extra virgin olive oil on cardiovascular risk factors: A systematic review and meta-analysis. Crit Rev Food Sci Nutr. 2019;59(17):2772-2795. doi: 10.1080/10408398.2018.1470491. Epub 2018 Nov 13. PMID 29708409
- [Background] Jimenez-Torres J, Alcala-Diaz JF, Torres-Pena JD, Gutierrez-Mariscal FM, Leon-Acuna A, Gomez-Luna P, Fernandez-Gandara C, Quintana-Navarro GM, Fernandez-Garcia JC, Perez-Martinez P, Ordovas JM, Delgado-Lista J, Yubero-Serrano EM, Lopez-Miranda J. Mediterranean Diet Reduces Atherosclerosis Progression in Coronary Heart Disease: An Analysis of the CORDIOPREV Randomized Controlled Trial. Stroke. 2021 Nov;52(11):3440-3449. doi: 10.1161/STROKEAHA.120.033214. Epub 2021 Aug 10. Erratum In: Stroke. 2021 Nov;52(11):e754. doi: 10.1161/STR.0000000000000393. PMID 34372670
- [Background] Patti AM, Carruba G, Cicero AFG, Banach M, Nikolic D, Giglio RV, Terranova A, Soresi M, Giannitrapani L, Montalto G, Stoian AP, Banerjee Y, Rizvi AA, Toth PP, Rizzo M. Daily Use of Extra Virgin Olive Oil with High Oleocanthal Concentration Reduced Body Weight, Waist Circumference, Alanine Transaminase, Inflammatory Cytokines and Hepatic Steatosis in Subjects with the Metabolic Syndrome: A 2-Month Intervention Study. Metabolites. 2020 Oct 2;10(10):392. doi: 10.3390/metabo10100392. PMID 33023123
- [Background] Gaforio JJ, Visioli F, Alarcon-de-la-Lastra C, Castaner O, Delgado-Rodriguez M, Fito M, Hernandez AF, Huertas JR, Martinez-Gonzalez MA, Menendez JA, Osada J, Papadaki A, Parron T, Pereira JE, Rosillo MA, Sanchez-Quesada C, Schwingshackl L, Toledo E, Tsatsakis AM. Virgin Olive Oil and Health: Summary of the III International Conference on Virgin Olive Oil and Health Consensus Report, JAEN (Spain) 2018. Nutrients. 2019 Sep 1;11(9):2039. doi: 10.3390/nu11092039. PMID 31480506
- [Background] Sayon-Orea C, Razquin C, Bullo M, Corella D, Fito M, Romaguera D, Vioque J, Alonso-Gomez AM, Warnberg J, Martinez JA, Serra-Majem L, Estruch R, Tinahones FJ, Lapetra J, Pinto X, Tur JA, Lopez-Miranda J, Bueno-Cavanillas A, Delgado-Rodriguez M, Matia-Martin P, Daimiel L, Sanchez VM, Vidal J, Vazquez C, Ros E, Ruiz-Canela M, Sorli JV, Castaner O, Fiol M, Navarrete-Munoz EM, Aros F, Gomez-Gracia E, Zulet MA, Sanchez-Villegas A, Casas R, Bernal-Lopez R, Santos-Lozano JM, Corbella E, Bouzas C, Garcia-Arellano A, Basora J, Asensio EM, Schroder H, Monino M, Garcia de la Hera M, Tojal-Sierra L, Toledo E, Diaz-Lopez A, Goday A, Salas-Salvado J, Martinez-Gonzalez MA. Effect of a Nutritional and Behavioral Intervention on Energy-Reduced Mediterranean Diet Adherence Among Patients With Metabolic Syndrome: Interim Analysis of the PREDIMED-Plus Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1486-1499. doi: 10.1001/jama.2019.14630. PMID 31613346
- [Background] Riboli E, Kaaks R. The EPIC Project: rationale and study design. European Prospective Investigation into Cancer and Nutrition. Int J Epidemiol. 1997;26 Suppl 1:S6-14. doi: 10.1093/ije/26.suppl_1.s6. PMID 9126529
- [Background] Jurado-Ruiz E, Varela LM, Luque A, Berna G, Cahuana G, Martinez-Force E, Gallego-Duran R, Soria B, de Roos B, Romero Gomez M, Martin F. An extra virgin olive oil rich diet intervention ameliorates the nonalcoholic steatohepatitis induced by a high-fat "Western-type" diet in mice. Mol Nutr Food Res. 2017 Mar;61(3). doi: 10.1002/mnfr.201600549. Epub 2016 Dec 13. PMID 27749006
- [Background] Saibandith B, Spencer JPE, Rowland IR, Commane DM. Olive Polyphenols and the Metabolic Syndrome. Molecules. 2017 Jun 29;22(7):1082. doi: 10.3390/molecules22071082. PMID 28661446
- [Background] Mirabelli M, Chiefari E, Arcidiacono B, Corigliano DM, Brunetti FS, Maggisano V, Russo D, Foti DP, Brunetti A. Mediterranean Diet Nutrients to Turn the Tide against Insulin Resistance and Related Diseases. Nutrients. 2020 Apr 12;12(4):1066. doi: 10.3390/nu12041066. PMID 32290535
- [Background] Yubero-Serrano EM, Lopez-Moreno J, Gomez-Delgado F, Lopez-Miranda J. Extra virgin olive oil: More than a healthy fat. Eur J Clin Nutr. 2019 Jul;72(Suppl 1):8-17. doi: 10.1038/s41430-018-0304-x. PMID 30487558